CLINICAL TRIAL: NCT02293109
Title: Phase I Study of Escalating Doses of Carfilzomib With Hyper-CVAD in Patients With Newly Diagnosed Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Carfilzomib and Hyper-CVAD in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mehrdad Abedi, MD (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Mehrdad Abedi, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 660258; UCDCC#246 (Registry Identifier: UC Davis); UCDCC#246 (Other: University of California Davis); NCI-2014-02245 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Contiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — carfilzomib; Cyclophosphamide; Vincristine; Doxorubicin; Dexamethasone; Calcium Dobesilate; Methotrexate; merphos; Cytarabine; Leucovorin; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carfilzomib and hyper-CVAD) (Experimental): Patients receive carfilzomib IV over 30 minutes on days 0, 1, 7, and 8. Patients also receive hyper-CVAD comprising cyclophosphamide IV over 2 hours every 12 hours for 6 doses beginning on day 1, vincristine sulfate IV on days 4 and 11, doxorubicin hydrochloride IV over 2-24 hours on day 4, and dexamethasone PO on days 1-4 and 11-14 (courses 1 and 3) and methotrexate IV over 24 hours on day 1, cytarabine IV over 2 hours every 12 hours for 4 doses starting on day 2, leucovorin calcium IV or PO every 6 hours beginning 36 hours after the start of methotrexate infusion, and methylprednisolone IV every 12 hours for 6 doses beginning on day 1 (courses 2 and 4). Patients with CD20 positive disease also receive rituximab twice daily on days 1 and 11 of courses 1 and 3 and days 1 and 8 of courses 2 and 4. Treatment repeats every 3-4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carfilzomib; Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: doxorubicin hydrochloride; Drug: dexamethasone; Drug: methotrexate; Drug: cytarabine; Drug: leucovorin calcium; Drug: methylprednisolone; Biological: rituximab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: leucovorin calcium — Given IV or PO
  Other Names: CF; CFR; LV
Drug: methylprednisolone — Given IV
  Other Names: Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort
Biological: rituximab
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of carfilzomib when given together with the hyperfractionated (hyper)-cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone (CVAD) chemotherapy regimen in treating patients with newly diagnosed acute lymphoblastic leukemia or lymphoma. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving carfilzomib with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Safety and tolerability of administering carfilzomib in combination with hyper-CVAD chemotherapy.

II. Recommended dose of carfilzomib in combination with hyper-CVAD chemotherapy for the future phase II trial.

SECONDARY OBJECTIVES:

I. Rate of remission after 2nd and 4th cycles. II. Incidence of minimal residual disease by flow cytometry at 4th cycle.

OUTLINE: This is a dose escalation study of carfilzomib.

Patients receive carfilzomib intravenously (IV) over 30 minutes on days 0, 1, 7, and 8. Patients also receive hyper-CVAD comprising cyclophosphamide IV over 2 hours every 12 hours for 6 doses beginning on day 1, vincristine sulfate IV on days 4 and 11, doxorubicin hydrochloride IV over 2-24 hours on day 4, and dexamethasone orally (PO) on days 1-4 and 11-14 (courses 1 and 3) and methotrexate IV over 24 hours on day 1, cytarabine IV over 2 hours every 12 hours for 4 doses starting on day 2, leucovorin calcium IV or PO every 6 hours beginning 36 hours after the start of methotrexate infusion, and methylprednisolone IV every 12 hours for 6 doses beginning on day 1 (courses 2 and 4). Patients with cluster of differentiation (CD)20 positive disease also receive rituximab twice daily on days 1 and 11 of courses 1 and 3 and days 1 and 8 of courses 2 and 4. Treatment repeats every 3-4 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Newly diagnosed acute lymphoblastic leukemia/lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (3 if it is directly disease related and is expected to get better if the acute lymphoblastic leukemia/lymphoma [ALL] is under control)
* Left ventricular ejection fraction (LVEF) > 40%
* Total bilirubin =< 3 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.5 x upper limit of normal
* Creatinine clearance (CrCl) >= 45 mL/minute within 7 days prior to enrollment either measured or calculated using a standard formula (eg, Cockcroft and Gault); in cases that creatinine clearance cannot be measured accurately, 24 hour urine can be used
* Disease free of other malignancies beside the ALL at the time of the study
* Male subjects must agree to practice contraception
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 24 hours prior to the initiation of the study and they must agree to ongoing pregnancy testing and to practice contraception

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females
* Active congestive heart failure (New York Heart Association [NYHA] class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention
* Unstable angina or myocardial infarction within 6 months prior to enrollment, NYHA class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities unless subject has a pacemaker
* Uncontrolled hypertension, uncontrolled pulmonary hypertension or uncontrolled diabetes within 14 days prior to enrollment
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 14 days of baseline
* Known history of allergy to Captisol®
* Known sero-positive for active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are sero-positive because of hepatitis B virus vaccine are eligible
* Breakpoint cluster region-Abelson positive (BCR-ABL +) patients will be excluded from the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of carfilzomib with hyper-CVAD, defined as the dose that produces dose limiting toxicity in 17% or fewer (1/6) of patients, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4 | Up to 56 days (after second course)
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by NCI CTCAE version 4.0) and nadir or maximum values for the laboratory measures, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.

SECONDARY OUTCOMES:
Rate of remission | Up to 56 days (after second course)
  All responses will be reported. Response rate among patients with measurable disease will be summarized by exact binomial confidence intervals.
Rate of minimal residual disease (MRD) in bone marrow aspirate samples | Up to 56 days (after second course)
  MRD will be defined an aberrant expression of at least 2 antigens in comparison with the known patterns of antigen expression by normal maturing CD19 positive B-cells. A distinct cluster of at least 20 cells showing altered antigen expression will be characterized as an aberrant cell population.
Rate of MRD in bone marrow aspirate samples | Up to 112 days (after 4th course)
  MRD will be defined an aberrant expression of at least 2 antigens in comparison with the known patterns of antigen expression by normal maturing CD19 positive B-cells. A distinct cluster of at least 20 cells showing altered antigen expression will be characterized as an aberrant cell population.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Abedi, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States